CLINICAL TRIAL: NCT06784180
Title: Intrathecal Hydromorphone vs Intrathecal Morphine to Treat Post Cesarean Pain in Patients With Opioid Use Disorder Taking Buprenorphine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-3302
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
Keywords: Morphine; Hydromorphone; Intrathecal; Suboxone; Opioid use disorder; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine; Bupivacaine; Fentanyl; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomly allocated to receive either 200 mcg of intrathecal morphine or 100 mcg of intrathecal hydromorphone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a single center, double-blind, randomized trial. The randomization process will occur through the use of a computer generated randomization scheme with allocation concealment in numbered opaque envelopes carried out by a blinded observer. Following randomization, opioid medications will be prepared by an anesthesia provider who is not involved in the clinical care of the patient. The opioid medications will be prepared so that the volume will be the same for both medications to ensure adequate blinding. Opioid medications will be either 200 mcg of preservative free morphine (0.4mL) or 100mcg of preservative free hydromorphone (0.1 mL) with 0.3 mL of saline added for a total volume of 0.4mL. The opioid medication will be labeled "intrathecal opioid" and given to the anesthesia provider that will be taking care of the patient. The anesthesia provider collecting the postoperative data will also be blinded to which intrathecal opioid medication the patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): Participants in this arm will receive intrathecal 200 mcg of preservative free morphine (0.4mL) with administration of 0.75% bupivacaine in 8.25% dextrose (dose determined by patient weight, height, gestational age) and 15 mcg fentanyl
  Interventions: Drug: Morphine; Drug: Bupivacaine; Drug: Fentanyl
- Intrathecal Hydromorphone (Experimental): Participants in this arm will receive intrathecal 100 mcg of preservative free hydromorphone (0.1mL) with 0.3mL of saline added for a total volume of 0.4mL with administration of 0.75% bupivacaine in 8.25% dextrose (dose determined by patient weight, height, gestational age) and 15 mcg fentanyl
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Drug: Hydromorphone

INTERVENTIONS:
Drug: Morphine — 200 mcg intrathecal morphine
  Other Names: Duramorph
  Arms: Intrathecal Morphine
Drug: Bupivacaine — Intrathecal 0.75% bupivacine in 8.25% dextrose (Dose determined by weight, height, gestational age)
  Other Names: Marcaine, Sensoricaine, Posimir
Drug: Fentanyl — 15 mcg intrathecal fentanyl
  Other Names: Duragesic, Subsys
Drug: Hydromorphone — 100 mcg intrathecal hydromorphone
  Other Names: Dilaudid, Exalgo
  Arms: Intrathecal Hydromorphone

SUMMARY:
This is a single center, double-blind, randomized trial to compare the effects of intrathecal hydromorphone versus intrathecal morphine to treat post cesarean pain in patients with OUD taking buprenorphine. Inclusion criteria include American Society of Anesthesiologists (ASA) Physical Status II or III presenting for cesarean delivery to be done under spinal anesthesia, who have a diagnosis of OUD and are taking buprenorphine. Exclusion criteria include contraindication to spinal anesthesia, allergy/intolerance to acetaminophen or ibuprofen and laboring patients who have an epidural that will be used for anesthesia for cesarean delivery. Potential subjects will be approached about participating in the study at either their preop anesthesia visit or on the day of surgery after surgical and anesthesia consent has been obtained. Enrolled patients will be randomly allocated to receive either 200 mcg of intrathecal morphine or 100 mcg of intrathecal hydromorphone (study opioid medication). Intraoperatively, with the patient in a sitting position a spinal block will be performed with administration of 0.75% bupivacaine in 8.25% dextrose, 15 mcg fentanyl and the study opioid medication. Supplemental intraoperative analgesia/anxiolysis will be administered at the discretion of the anesthesia care team. Ultrasound-guided transversus abdominis plane blocks will be performed bilaterally at the end of the procedure with 10mL liposomal bupivacaine mixed with 10mL 0.25% bupivacaine injected on each side. Post-cesarean multimodal pain regimen will include scheduled acetaminophen 650mg every 6 hours and scheduled ibuprofen 600mg every 6 hours. Oxycodone will be ordered for breakthrough pain, starting at 5mg every 6 hours as needed. Escalation of as needed pain medication will be at the discretion of the anesthesia team. The patient will be followed for the following 36 hours postoperatively. The primary outcome is the patient's pain score with movement at 12 hours. Secondary outcomes include pain scores at rest and with movement at 6 and 24 hours, satisfaction with anesthesia, time to first opioid use, total opioid consumption in 24 and 36 hours, subjective rating of nausea and pruritis over first 24 hours , treatment for nausea or pruritis in 24 and 36 hours, Obstetric Quality of Recovery 10 (ObsQoR10) score, and Global Health Numeric Rating Scale (NRS) score.

DETAILED DESCRIPTION:
Background:

Opioid use disorder (OUD) and neonatal abstinence syndrome (NAS) has increased significantly in pregnancy during the last decade. Lui et al found the rate of OUD in patients undergoing cesarean delivery increased 4 fold from 2007 to 2014. Untreated addiction can lead to increased risk of preterm birth, low birth weight and fetal death. Women with OUD were at higher risk for inpatient mortality and readmission following delivery, particularly those who had a cesarean delivery. Pregnancy outcomes are improved if women with OUD are treated with opioid agonist therapy during pregnancy. The American College of Obstetricians and Gynecologists recommends universal screening for substance use during pregnancy, and initiation of medication assisted treatment (MAT) with opioid agonist therapy. The most commonly used MATs are methadone and buprenorphine. Methadone, a full opioid agonist, is only dispensed via federally regulated opioid treatment programs and requires patients to present daily for their methadone treatment. Buprenorphine, a partial opioid agonist, can be prescribed by a physician and patients are able to treat themselves at home. Because buprenorphine is more easily dispensed, more patients are treated with buprenorphine for OUD.

Continuation of MAT is recommended during the peripartum period to help prevent relapse post-partum. Managing pain for parturients on MAT for OUD can be challenging, particularly for patients taking buprenorphine because of its ability to compete with other opioids at the mu receptor. Women delivering via cesarean who are taking buprenorphine for MAT generally have higher postop opioid use compared to women without OUD. This was particularly true for the immediate 24 hour postop period. A recent collaboration publication between the Society for Obstetric Anesthesiology and Perinatology and Society for Maternal Fetal Medicine highlights the lack of quality research on peripartum pain management in the OUD population.

Various strategies to improve postop pain management in this patient population have been used. Use of continuous epidural infusions postop does improve pain control but has the disadvantage of resulting in weakness that can limit mobility. Others have used low dose ketamine for management of post-cesarean pain. Use of intrathecal (IT) clonidine showed some benefit, however they have higher risk for intra- and postoperative hypotension. Continuous epidural or IV infusions tend to limit patients' functionality postop due to need to be physically connected to a device to receive these treatments.

Buprenorphine is a partial agonist at the mu opioid receptor and therefore has low activity. However, it has very high binding affinity for the mu opioid receptor making it very competitive with other opioid agonists. Hydromorphone also has high binding affinity for the mu opioid receptor, allowing it to more effectively compete for binding in the presence of buprenorphine. Morphine has lower binding affinity at the mu opioid receptor making it less able to compete with buprenorphine.

A multisociety expert panel recommends continuation of buprenorphine therapy in the perioperative period, noting that studies have shown that adequate analgesia can be achieved and relapse potential is higher when buprenorphine is discontinued. They recommend nonopioid strategies for pain management, including use of regional anesthesia, NSAIDs and acetaminophen.

Inclusion of IT long-acting opioid with spinal anesthesia is considered standard of care for post-cesarean pain management. Traditionally IT morphine has been used but more recent studies have looked at use of IT hydromorphone instead of IT morphine. A retrospective study comparing 0.1mg IT morphine to 0.04mg IT hydromorphone found no difference in 24 hour pain scores or 24 hour total opioid consumption. While Marroquin et al found a shorter interval to first opioid use and higher total opioid consumption in the IT hydromorphone group compared to the IT morphine group, they still concluded that hydromorphone was a reasonable alternative to morphine. Sharpe et al showed no difference in pain scores or postop opioid consumption in patients receiving IT hydromorphone compared to morphine. This study excluded patients with history of chronic pain syndromes. These studies demonstrate IT hydromorphone is a safe and effective alternative to IT morphine. Because of the pharmacological properties of buprenorphine, hydromorphone and morphine the investigators hypothesize that the use of IT hydromorphone will provide superior pain control to IT morphine in the presence of buprenorphine.

Methods:

This will be a single center, double-blind, randomized trial to compare the effects of IT hydromorphone vs morphine to treat post cesarean pain in patients with OUD taking buprenorphine. Inclusion criteria include American Society of Anesthesiologists (ASA) Physical Status II or III presenting for cesarean delivery to be done under spinal anesthesia, who have a diagnosis of OUD and are taking buprenorphine. Exclusion criteria include contraindication to spinal anesthesia, allergy/intolerance to acetaminophen or ibuprofen and laboring patients who have an epidural that will be used for anesthesia for cesarean delivery.

Potential subjects will be approached about participating in the study at either their preop anesthesia visit or on the day of surgery after surgical and anesthesia consent has been obtained. Only licensed physician investigators will recruit patients and written informed consent will be obtained. No remuneration will be provided.

The randomization process will occur through use of a computer generated randomization scheme with allocation concealment in numbered opaque envelopes carried out by a blinded observer. Enrolled patients will be randomly allocated to receive either 200 mcg of IT morphine or 100 mcg of IT hydromorphone. Following randomization, opioid medications will be prepared by an anesthesia provider who is not involved in the clinical care of the patient. The opioid medications will be prepared so that the volume will be the same for both medications to ensure adequate blinding. Opioid medications will be either 200mcg of preservative free morphine (0.4mL) or 100mcg of preservative free hydromorphone (0.1mL) with 0.3mL of saline added for a total volume of 0.4mL. The opioid medication will be labeled "intrathecal opioid" and given to the anesthesia provider that will be taking care of the patient.

Patients will be brought to the operating room on labor and delivery where standard ASA monitors will be applied and an IV fluid co-load with lactated ringers will be started. With the patient in a sitting position a spinal block will be performed with administration of 0.75% bupivacaine in 8.25% dextrose, 15 mcg fentanyl and the study opioid medication. The patient will then be placed in the supine position and an infusion of phenylephrine will be started and titrated to maintain baseline blood pressure, as is our standard protocol. All patients will receive ondansetron and dexamethasone for antiemetic prophylaxis. Additional antiemetics will be administered as needed to treat intraoperative nausea. After delivery, oxytocin will be administered per institutional protocol. Supplemental intraoperative analgesia/anxiolysis will be administered at the discretion of the anesthesia care team. Ultrasound-guided transversus abdominis plane blocks will be performed bilaterally at the end of the procedure with 10mL liposomal bupivacaine mixed with 10mL 0.25% bupivacaine injected on each side. Respiratory rate and sedation will be assessed every 2 hours for 12 hours by nursing staff. Naloxone 0.4 mg will be administered for respiratory rate <6 or if patient is unarousable. All post-cesarean pain needs are managed by the anesthesia team at UNC. Post-cesarean multimodal pain regimen will include scheduled acetaminophen 650mg every 6 hours and scheduled ibuprofen 600mg every 6 hours. Oxycodone will be ordered for breakthrough pain, starting at 5mg every 6 hours as needed. Escalation of as needed pain medication will be at the discretion of the anesthesia team. Ondansetron and promethazine will be ordered to treat nausea as needed. Treatment of opioid induced pruritus with nalbuphine or naloxone will be at the discretion of the anesthesia care team in collaboration with the patient.

Early end points: Change in fetal or maternal health mandating the use of other anesthetic techniques, inability to perform the spinal technique, withdrawal of subject consent at any time

Surgical complications resulting in the need for additional surgical procedures: There will be no additional costs to the patient as a result of participation in this study. The costs of routine labor and delivery analgesia and anesthetic care will be the responsibility of the patient and their insurance provider.

Risks and Discomforts:

Hypotension is one of the most common sequelae from spinal anesthesia techniques. Intravascular volume expansion and standardized vasopressor treatment will be immediately available and utilized as needed. The risk of hypotension will not be increased due to the randomization of study medications.

Approximately 10-40% of the time, nausea may occur during a cesarean delivery. If nausea occurs, it will be treated and managed according to usual measures. Approximately 10% of the time pruritus may occur, which will be treated and managed according to usual measures.

The risk of a post dural puncture headache (PDPH) exists for spinal techniques. The risk is approximately 1% in an obstetric population with a 25 gauge Whitacre needle, and will not be increased by the administration of study medications. If a PDPH occurs, various methods are available for treatment and will be discussed with the patient.

Uncommon (less than 1%) sequelae include failure to obtain anesthesia, incomplete anesthesia, and need to repeat the spinal anesthetic. There is less than 0.1% risk of infection, epidural or spinal hematomas, and nerve injury. The use of the study medications will not increase these risks.

Potential Benefits: Patients may experience improved pain control with fewer opioid related side effects. Information from this study may benefit other patients undergoing neuraxial anesthesia for cesarean delivery.

Assurance of safety and tolerability:

Following continuous care during the cesarean delivery, all patients will have a scheduled visit with study personnel at 6, 12 and 24 hours after IT injection to evaluate the efficacy of analgesia. As noted, numerical rating scale pain scores, satisfaction, and opioid side effects will be recorded. Patients will also be evaluated for pain by nursing staff per unit protocol.

A patient may withdraw from the study at any time.

Serious Adverse Experiences: Any serious or unexpected adverse experiences, whether or not considered to be related to the study, shall be reported immediately via the UNC patient safety reporting system. These events are reviewed by the Director of Obstetric Anesthesia. Anyone involved in the patients' care will be able to report adverse experiences.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status II or III presenting for cesarean delivery to be done under spinal anesthesia,
* have a diagnosis of OUD
* taking buprenorphine

Exclusion Criteria:

* Contraindication to spinal anesthesia,
* allergy/intolerance to acetaminophen or ibuprofen
* laboring patients who have an epidural that will be used for anesthesia for cesarean delivery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pain score with movement | 12 hours postoperatively
  Using the pain rating scale, patient will score pain with movement (1-10, 10 being worst pain) at 12 hours postoperatively

SECONDARY OUTCOMES:
Pain scores at rest | 6 and 24 hours postoperatively
  Using the pain rating scale, patient will score pain at rest (1-10, 10 being worst pain) at 6 and 24 hours postoperatively
Pain with movement | 6 and 24 hours postoperatively
  Using the pain rating scale, patient will score pain with movement (1-10, 10 being worst pain) at 6 and 24 hours postoperatively
Satisfaction with anesthesia | Within 24 hours postoperatively
  Overall satisfaction with analgesia: 4 = satisfied, 3 = somewhat satisfied, 2 = neutral, 1 = somewhat dissatisfied, 0 = dissatisfied
Time to first opioid use | Within 72 hours postoperatively
  Time at which the patient has first dose of systemic opioid pain medication postoperatively within 72 hours
Total opioid consumption | 24 and 36 hours postoperatively
  Total opioids (converted into morphine mg equivalents) in 24 and 36 hours postoperatively
Subjective rating of nausea and pruritus | Over first 24 hours postoperatively
  Patient subjective assessment of nausea and pruritus in first 24 hours postoperatively: 0 = none, 1 = mild, 2 = moderate, 3 = severe
Treatment for nausea | 24 and 36 hours postoperatively
  Chart review of number of enrolled patients who required treatment for nausea (antiemetics). This will be reported as x participants/46 total participants (%) were treated for nausea at 24 and 36 hours postoperatively
Treatment for pruritus | 24 and 36 hours postoperatively
  Chart review of number of enrolled patients who required treatment for pruritus (nalbuphine or naloxone). This will be reported as x participants/46 total participants (%) were treated for pruritus at 24 and 36 hours postoperatively
Obstetric Quality of Recovery 10 (ObsQoR10) score | 24 hours postoperatively
  10 total questions
  Measures pain, nausea/vomiting, dizziness with scale 0-10 (0 meaning no pain, 10 meaning worst imaginable pain), higher score means worse outcome
  Measures patient comfort, and ability to independently mobilize, hold baby without assistance, feed/nurse baby without assistance, look after personal hygiene/toilet, and overall sense of patient control with scale 0-10 (0 meaning no/never, 10 meaning yes/always), higher score means better outcome
Global Health Numeric Rating Scale (NRS) score | 24 hours postoperatively
  1 total question
  Measures pain over the past 24 hours postoperatively with scale 0-100 (0 meaning worst imaginable pain, and 100 meaning no pain)
  Higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amy Penwarden, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Hirai AH, Ko JY, Owens PL, Stocks C, Patrick SW. Neonatal Abstinence Syndrome and Maternal Opioid-Related Diagnoses in the US, 2010-2017. JAMA. 2021 Jan 12;325(2):146-155. doi: 10.1001/jama.2020.24991. PMID 33433576
- [Background] Lui B, Aaronson JA, Tangel V, Quincy M, Weinberg R, Abramovitz SE, White RS. Opioid use disorder and maternal outcomes following cesarean delivery: a multistate analysis, 2007-2014. J Comp Eff Res. 2020 Jul;9(10):667-677. doi: 10.2217/cer-2020-0050. Epub 2020 Jul 10. PMID 32648478
- [Background] Suarez EA, Huybrechts KF, Straub L, Hernandez-Diaz S, Jones HE, Connery HS, Davis JM, Gray KJ, Lester B, Terplan M, Mogun H, Bateman BT. Buprenorphine versus Methadone for Opioid Use Disorder in Pregnancy. N Engl J Med. 2022 Dec 1;387(22):2033-2044. doi: 10.1056/NEJMoa2203318. PMID 36449419
- [Background] Vilkins AL, Bagley SM, Hahn KA, Rojas-Miguez F, Wachman EM, Saia K, Alford DP. Comparison of Post-Cesarean Section Opioid Analgesic Requirements in Women With Opioid Use Disorder Treated With Methadone or Buprenorphine. J Addict Med. 2017 Sep/Oct;11(5):397-401. doi: 10.1097/ADM.0000000000000339. PMID 28727661
- [Background] Mittal L, Suzuki J. Feasibility of collaborative care treatment of opioid use disorders with buprenorphine during pregnancy. Subst Abus. 2017 Jul-Sep;38(3):261-264. doi: 10.1080/08897077.2015.1129525. Epub 2015 Dec 16. PMID 26672650
- [Background] Cobb J, Craig W, Richard J, Snow E, Turcotte H, Warters R, Quaye A. A Retrospective Study of Acute Postoperative Pain After Cesarean Delivery in Patients With Opioid Use Disorder Treated With Opioid Agonist Pharmacotherapy. J Addict Med. 2022 Sep-Oct 01;16(5):549-556. doi: 10.1097/ADM.0000000000000964. Epub 2022 Feb 14. PMID 35165223
- [Background] Meyer M, Paranya G, Keefer Norris A, Howard D. Intrapartum and postpartum analgesia for women maintained on buprenorphine during pregnancy. Eur J Pain. 2010 Oct;14(9):939-43. doi: 10.1016/j.ejpain.2010.03.002. Epub 2010 May 4. PMID 20444630
- [Background] Holland E, Gibbs L, Spence NZ, Young M, Werler MM, Guang Z, Saia K, Bateman BT, Achu R, Wachman EM. A comparison of postpartum opioid consumption and opioid discharge prescriptions among opioid-naive patients and those with opioid use disorder. Am J Obstet Gynecol MFM. 2023 Aug;5(8):101025. doi: 10.1016/j.ajogmf.2023.101025. Epub 2023 May 19. PMID 37211090
- [Background] O'Connor AB, Smith J, O'Brien LM, Lamarche K, Byers N, Nichols SD. Peripartum and Postpartum Analgesia and Pain in Women Prescribed Buprenorphine for Opioid Use Disorder Who Deliver by Cesarean Section. Subst Abuse. 2022 Jun 21;16:11782218221107936. doi: 10.1177/11782218221107936. eCollection 2022. PMID 35754980
- [Background] Reno JL, Kushelev M, Coffman JH, Prasad MR, Meyer AM, Carpenter KM, Palettas MS, Coffman JC. Post-Cesarean Delivery Analgesic Outcomes in Patients Maintained on Methadone and Buprenorphine: A Retrospective Investigation. J Pain Res. 2020 Dec 30;13:3513-3524. doi: 10.2147/JPR.S284874. eCollection 2020. PMID 33408510
- [Background] Lim G, Soens M, Wanaselja A, Chyan A, Carvalho B, Landau R, George RB, Klem ML, Osmundson SS, Krans EE, Terplan M, Bateman BT. A Systematic Scoping Review of Peridelivery Pain Management for Pregnant People With Opioid Use Disorder: From the Society for Obstetric Anesthesia and Perinatology and Society for Maternal Fetal Medicine. Anesth Analg. 2022 Nov 1;135(5):912-925. doi: 10.1213/ANE.0000000000006167. Epub 2022 Sep 22. PMID 36135926
- [Background] Stanislaus MA, Reno JL, Small RH, Coffman JH, Prasad M, Meyer AM, Carpenter KM, Coffman JC. Continuous Epidural Hydromorphone Infusion for Post-Cesarean Delivery Analgesia in a Patient on Methadone Maintenance Therapy: A Case Report. J Pain Res. 2020 Apr 28;13:837-842. doi: 10.2147/JPR.S242271. eCollection 2020. PMID 32425588
- [Background] Cobb J, Craig W, Richard J, Snow E, Turcotte H, Warters R, Quaye A. Low-dose ketamine infusion for post-cesarean delivery analgesia in patients with opioid use disorder. Int J Obstet Anesth. 2021 Aug;47:103170. doi: 10.1016/j.ijoa.2021.103170. Epub 2021 May 2. No abstract available. PMID 34090769
- [Background] Cook MI, Kushelev M, Coffman JH, Coffman JC. Analgesic Outcomes in Opioid Use Disorder Patients Receiving Spinal Anesthesia with or without Intrathecal Clonidine for Cesarean Delivery: A Retrospective Investigation. J Pain Res. 2022 Apr 21;15:1191-1201. doi: 10.2147/JPR.S358045. eCollection 2022. PMID 35478995
- [Background] Volpe DA, McMahon Tobin GA, Mellon RD, Katki AG, Parker RJ, Colatsky T, Kropp TJ, Verbois SL. Uniform assessment and ranking of opioid mu receptor binding constants for selected opioid drugs. Regul Toxicol Pharmacol. 2011 Apr;59(3):385-90. doi: 10.1016/j.yrtph.2010.12.007. Epub 2011 Jan 6. PMID 21215785
- [Background] Kohan L, Potru S, Barreveld AM, Sprintz M, Lane O, Aryal A, Emerick T, Dopp A, Chhay S, Viscusi E. Buprenorphine management in the perioperative period: educational review and recommendations from a multisociety expert panel. Reg Anesth Pain Med. 2021 Oct;46(10):840-859. doi: 10.1136/rapm-2021-103007. Epub 2021 Aug 12. PMID 34385292
- [Background] Beatty NC, Arendt KW, Niesen AD, Wittwer ED, Jacob AK. Analgesia after Cesarean delivery: a retrospective comparison of intrathecal hydromorphone and morphine. J Clin Anesth. 2013 Aug;25(5):379-383. doi: 10.1016/j.jclinane.2013.01.014. Epub 2013 Aug 17. PMID 23965210
- [Background] Marroquin B, Feng C, Balofsky A, Edwards K, Iqbal A, Kanel J, Jackson M, Newton M, Rothstein D, Wong E, Wissler R. Neuraxial opioids for post-cesarean delivery analgesia: can hydromorphone replace morphine? A retrospective study. Int J Obstet Anesth. 2017 May;30:16-22. doi: 10.1016/j.ijoa.2016.12.008. Epub 2016 Dec 30. PMID 28185794
- [Background] Sharpe EE, Molitor RJ, Arendt KW, Torbenson VE, Olsen DA, Johnson RL, Schroeder DR, Jacob AK, Niesen AD, Sviggum HP. Intrathecal Morphine versus Intrathecal Hydromorphone for Analgesia after Cesarean Delivery: A Randomized Clinical Trial. Anesthesiology. 2020 Jun;132(6):1382-1391. doi: 10.1097/ALN.0000000000003283. PMID 32251031
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873